CLINICAL TRIAL: NCT04044183
Title: Active Brains: Managing Pain and Cognitions in Older Adults With Mild Cognitive Impairment (MCI) or Memory Related Problems (MRP) and Chronic Pain
Brief Title: Managing Pain and Cognitions in Older Adults With Mild Cognitive Impairment or Memory Related Problems and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Associate Professor/Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P002152
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain; Mild Cognitive Impairment; Older Adults; Physical Activity
Keywords: Chronic Pain; Mild Cognitive Impairment; Older Adults; Physical Activity; Memory Related Problems
MeSH Terms: conditions — Chronic Pain; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Brains (Experimental): Active Brains uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions, and weekly practice assignments (homework). The Active Brains sessions reflect a purposeful integration of the three treatment approaches (relaxation methods, stress appraisal & coping, and growth enhancement). The format is an 8-week program with weekly meetings and a focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. Active Brains 1 uses a digital monitoring device (i.e., Fitbit) for recording of physical activity.
  Interventions: Behavioral: Active Brains 1; Behavioral: Active Brains 2
- Active Brains 2 (Placebo Comparator): This active comparison condition controls for the effect of time spent, group member support/feedback, and interventionist support/feedback. The original HEP was adapted to provide population-specific information on chronic pain and MCI/MRP symptoms. Participants also receive lifestyle education consistent from public health recommendations and standards for health promotion (e.g., "Sleep", "Nutrition", "Healthy Weight", and "Medical appointments"). The HEP program consists on 8 group sessions (each session is 90 minutes) that occur concurrently with the active intervention condition. The HEP is conducted in the same format as Active Brains-Fitbit but are not taught the mind-body, walking, or cognitive-behavioral skills. HEP participants are encouraged to set lifestyle goals instead of quota-based walking goals aided by the Fitbit as in the Active Brains-Fitbit condition.
  Interventions: Behavioral: Active Brains 1; Behavioral: Active Brains 2

INTERVENTIONS:
Behavioral: Active Brains 1 — Active Brains uses a multimodal approach to introduce and reinforce new skills, including didactics, in-session activities, discussions, and weekly practice assignments (homework). The Active Brains sessions reflect a purposeful integration of the three treatment approaches (relaxation methods, stress appraisal & coping, and growth enhancement). The format is an 8-week program with weekly meetings and a focus on relaxation response strategies, cognitive behavioral training, positive psychology and mind-body interactions. Active Brains 1 uses a digital monitoring device (i.e., Fitbit) for recording of physical activity.
Behavioral: Active Brains 2 — This active comparison condition controls for the effect of time spent, group member support/feedback, and interventionist support/feedback. The original HEP was adapted to provide population-specific information on chronic pain and MCI/MRP symptoms. Participants also receive lifestyle education consistent from public health recommendations and standards for health promotion (e.g., "Sleep", "Nutrition", "Healthy Weight", and "Medical appointments"). The HEP program consists on 8 group sessions (each session is 90 minutes) that occur concurrently with the active intervention condition. The HEP is conducted in the same format as Active Brains-Fitbit but are not taught the mind-body, walking, or cognitive-behavioral skills. HEP participants are encouraged to set lifestyle goals instead of quota-based walking goals aided by the Fitbit as in the Active Brains-Fitbit condition.

SUMMARY:
We aim to conduct a pilot randomized controlled trial comparing 2 symptom management programs for older adults with self-reported memory problems and chronic pain, Active Brains 1 and Active Brains 2. We will assess how each program may help in improving coping with pain and coping with cognitive functioning. We will explore feasibility, acceptability, and credibility and within group changes in physical, emotional and cognitive functioning.

DETAILED DESCRIPTION:
We aim to conduct a pilot randomized controlled trial comparing 2 symptom management programs for older adults with self-reported memory problems and chronic pain: Active Brains 1 Active Brains 2. We will assess how each program may help in improving coping with pain and coping with cognitive functioning. We will explore feasibility, acceptability, and credibility and within group changes in physical, emotional and cognitive functioning.

Each group meets for 8 90 minute sessions over a secure video platform. Each group has 5-8 participants. Participants receive a treatment manual. There are 2 assessment points: baseline, and post program. Assessments involve questionnaires, a walk test, and objective step count with ActiGraphs for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 60 years or older
* Have nonmalignant chronic pain for more than 3 months
* Has MCI or subjective memory related problems
* Able to perform a 6-minute walk test at an accelerated pace
* Owns a smartphone with Bluetooth 4.0
* Willingness and ability to participate in the Active Brains intervention and to comply with the requirements of the study protocol (including weekly sessions and Fitbit use)
* Free of concurrent psychotropic or pain medication for at least 2 weeks prior to initiation of treatment, OR stable on current psychotropic or pain medication for a minimum of 6 weeks and willing to maintain a stable dose
* Cleared by a medical doctor for study participation
* Leads a sedentary lifestyle

Exclusion Criteria:

* Diagnosed with medical illness expected to worsen in the next 6 months
* Serious mental illness or instability for which hospitalization may be likely in the next 6 months
* Current suicidal ideation reported on self-report
* Lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, or substance dependence
* Current substance use disorder, within the past 6 months
* Practice of yoga/meditation, or other mind-body techniques that elicit the relaxation response, once per week for 45 minutes or more within the last 3 months or less
* Regular use of Fitbit in the last 3 months
* Engagement in regular intensive physical exercise for >30 minute daily
* Unable to walk without use of assistance (e.g., wheelchair, walker)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doorley JD, Mace RA, Popok PJ, Grunberg VA, Ragnhildstveit A, Vranceanu AM. Feasibility Randomized Controlled Trial of a Mind-Body Activity Program for Older Adults With Chronic Pain and Cognitive Decline: The Virtual "Active Brains" Study. Gerontologist. 2022 Aug 12;62(7):1082-1094. doi: 10.1093/geront/gnab135. PMID 34487167
- [Derived] Mace RA, Doorley JD, Popok PJ, Vranceanu AM. Live Video Adaptations to a Mind-Body Activity Program for Chronic Pain and Cognitive Decline: Protocol for the Virtual Active Brains Study. JMIR Res Protoc. 2021 Jan 4;10(1):e25351. doi: 10.2196/25351. PMID 33208301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Brains | Active Brains 2
Started | 10 | 11
Completed | 8 | 11
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: While only 8 participants completed the Active Brains intervention, demographic data were available for all 9 participants who completed the baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Brains | Active Brains 2 | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (5.9) | 70.8 (8.4) | 69.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 10 | 17
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 11 | 20
Marital Status [Count of Participants; unit: Participants]
  Single, never married | 0 | 1 | 1
  Living with significant other | 3 | 6 | 9
  Married | 1 | 0 | 1
  Separated/Divorced | 2 | 3 | 5
  Widowed | 3 | 1 | 4
Education [Count of Participants; unit: Participants]
  Completed high school or GED (12 years) | 0 | 1 | 1
  Some college/Associates degree (<16 years) | 3 | 3 | 6
  Completed college (16 years) | 3 | 2 | 5
  Graduate/professional degree (>16 years) | 3 | 5 | 8
Employment [Count of Participants; unit: Participants]
  Employed full-time | 0 | 1 | 1
  Employed part-time | 1 | 1 | 2
  Retired | 4 | 6 | 10
  Unemployed | 1 | 1 | 2
  Other situation | 3 | 2 | 5
Pain medications [Count of Participants; unit: Participants]
  Opioids | 2 | 4 | 6
  Other analgesics | 5 | 4 | 9
  None | 2 | 3 | 5
Reported pain location [Count of Participants; unit: Participants]
  Upper | 3 | 4 | 7
  Lower | 2 | 0 | 2
  Multi-site | 4 | 7 | 11
Pain duration [Count of Participants; unit: Participants]
  Less than or equal to 5 years | 4 | 2 | 6
  6-10 years | 2 | 3 | 5
  Greater than or equal to 11 years | 3 | 6 | 9
Cognitive status [Count of Participants; unit: Participants]
  Normal | 4 | 8 | 12
  Cognitive Impairment | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire 3-Item (CSQ-3): Number of Participants With Scores Above and Below Scale Midpoint
Description: Items are summed to generate a total score; scores range from 3 to 12, with higher values indicating higher satisfaction
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants
  Scored above the scale midpoint | 8 | 9
  Scored below the scale midpoint | 0 | 1
  Did not complete the scale | 1 | 1

2. Secondary Outcome: Proportion of Participants With Valid Digital Monitoring Device Wear
Description: The proportion of patients with valid ActiGraph (digital monitoring device) wear for greater than or equal to 6 days (7+ hr/day) at baseline and 5 days at post test
Time Frame: 0 Weeks, 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants
  Wore the FitBit for at least 5 out of 7 days for 6 out of the 8 weeks of the program | 8 | 0
  Did not wear the FitBit for at least 5 out of 7 days for 6 out of the 8 weeks of the program | 1 | 11

3. Secondary Outcome: Proportion of Participants With Valid Adherence to Homework
Description: Proportion of participants completing at least 5 out of 7 days of homework assigned throughout the study
Time Frame: 0 Weeks, 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants
  Completed ≥ 5 of seven homework logs | 8 | 0
  Did not complete ≥ 5 of seven homework logs | 1 | 11

4. Secondary Outcome: Rate of Interventionist's Delivering the Programs by Following the Established Session Topics and Skills
Description: Percentage of audio recordings, progress notes, and checklists that were completed with 100% of content delivered for each session
Time Frame: 0 Weeks, 8 Weeks
Measure: Number; unit: percentage of therapist adherence
Units Other Than Participants: Sessions
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Number analyzed (Sessions) | 8 | 8
percentage of therapist adherence | 97.3 | 91.4

5. Secondary Outcome: Percentage of Missing or Low Reliability Measures (Feasibility of Quantitative Measures)
Description: Percentage of questionnaires that were entirely missing in >25% of participants and/or had an internal reliability below .70
Time Frame: 0 Weeks, 8 Weeks
Measure: Number; unit: Percentage of questionnaires were entire
Units Other Than Participants: Questionnaires
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Number analyzed (Questionnaires) | 19 | 19
Percentage of questionnaires were entire | 85 | 99

6. Secondary Outcome: Proportion of Participants Using Rescue (Non-Narcotic) Analgesics
Description: Single-item question on demographics form indicating whether participant used rescue (non-narcotic) analgesics at baseline
Time Frame: 0 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants | 4 | 5

7. Secondary Outcome: Proportion of Participants Using Narcotic Analgesics
Description: Single-item question on demographics form indicating whether participant used narcotic analgesics at baseline
Time Frame: 0 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants | 2 | 4

8. Secondary Outcome: Credibility and Expectancy Questionnaire (CEQ): Number of Participants With Scores Above and Below Scale Midpoint
Description: Number of participants rating expectations and believed credibility for the program above and below the scale midpoint, with higher ratings indicating more belief that the program is logical and will help with the intended outcome
Time Frame: 0 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
Participants
  Credibility: Scored above the scale midpoint | 9 | 11
  Credibility: Scored below the scale midpoint | 0 | 0
  Expectancy: Scored above the scale midpoint | 5 | 4
  Expectancy: Scored below the scale midpoint | 4 | 7

9. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: Assesses several cognitive domains and detection of mild cognitive impairment (MCI), with scores ranging from 0-30 and lower scores indicating greater cognitive decline
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 24.8 (2.4) | 26.3 (3.5)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 26.2 (1.7) | 26.6 (3.7)

10. Secondary Outcome: Godin Leisure-Time Exercise Questionnaire
Description: Rate of participant's leisure time and physical activity levels by indicating how many days per week are spent doing the activity for more than 15 minutes. Scores range from 0-119, with higher scores indicating greater levels of activity.
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 36 (34.9) | 20 (20.9)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 74 (57.5) | 30.8 (35.8)

11. Secondary Outcome: Measure of Current Status (MOCS-A)
Description: Rate of a participant's self-reported perceived stress self-management skills, with items ranging from 0-4 and a total score ranging from 0-52, and higher scores reflecting more usage of stress self-management skills
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 30.4 (12.4) | 25.6 (10.1)
  Post-Test: number analyzed (Participants) | 7 | 11
  Post-Test | 36.1 (14.2) | 28.3 (8.7)

12. Secondary Outcome: The Measurement of Everyday Cognition (eCog)
Description: Rate of participant's cognitively mediated functional abilities, with items ranging from 1-5. Total scores are an average of the items (range = 1-5), with higher scores indicating greater cognitive decline.
Time Frame: 0 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: mean of items
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 8 | 11
mean of items
  Baseline | 2.3 (1) | 1.9 (0.6)
  Post-Test | 2 (0.9) | 1.8 (0.5)

13. Secondary Outcome: Numerical Rating Scale
Description: Rate of a participant's pain at rest and with activity using a Likert scale with 0 being no pain and 10 being the worst possible pain
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Pain at rest (Baseline) | 5.9 (2.5) | 4.4 (2.6)
  Pain at rest (Post-Test): number analyzed (Participants) | 8 | 11
  Pain at rest (Post-Test) | 3.9 (2.1) | 4.3 (1.8)
  Pain with activity (Baseline) | 6.2 (1.8) | 5.7 (2.6)
  Pain with activity (Post-Test): number analyzed (Participants) | 8 | 11
  Pain with activity (Post-Test) | 4.2 (2.5) | 5.7 (2.2)

14. Secondary Outcome: The Cognitive and Affective Mindfulness Scale - Revised (CAMS-R)
Description: Rate of a participant's broad conceptualization of mindfulness, items range from 1-4 and scores range from 12-48, with higher values reflecting higher levels of mindfulness
Time Frame: 0 Weeks, 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 8 | 11
score on a scale
  Baseline | 31.9 (7.3) | 33.8 (8)
  Post-Test | 33.9 (6.1) | 35.3 (6)

15. Secondary Outcome: WHO Disability Assessment Schedule 2.0
Description: Rate of a participant's health and disability, with items ranging from 0-4, total scores ranging from 0-100, and higher scores reflecting greater disability
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 10 | 11
score on a scale
  Baseline | 17.1 (14.3) | 23.9 (17.2)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 16 (14.7) | 22.2 (15)

16. Secondary Outcome: The Gratitude Questionnaire (GQ-6)
Description: Rate of a participant's proneness to experience gratitude in daily life, with items ranging from 1-7, total scores ranging from 6-24, and a higher score indicating greater amount of gratitude
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 36.2 (5.9) | 32.5 (7.6)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 35.5 (7.1) | 35.9 (5.1)

17. Secondary Outcome: PROMIS Physical Function
Description: Rate of a participant's capability rather than performance of physical activities, with items ranging from 1-4, and total scores ranging from 8-40, with a higher score reflecting greater physical function
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 39.9 (5.5) | 37.1 (6.2)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 43.4 (9.6) | 38.2 (5.8)

18. Secondary Outcome: PROMIS Emotional Support
Description: Rate of a participant's perceived feelings of being cared and values for as an individual, with items ranging from 1-5. Items are normed to T-scores (mean = 50, standard deviation = 10), with higher T-scores indicating higher perceived social support.
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 51.1 (11.2) | 49.4 (9.6)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 52.1 (9.1) | 48.8 (9.5)

19. Secondary Outcome: T-Score for PROMIS Depression
Description: Rate of a participant's depressive symptoms, with items ranging from 1-5. Items are normed to T-scores (mean = 50, standard deviation = 10), with higher T-scores indicating higher depression.
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
T-score
  Baseline | 51.6 (6.6) | 55.6 (11.1)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 52.5 (8.6) | 54.3 (11.7)

20. Secondary Outcome: T-Score for PROMIS Anxiety
Description: Rate of a participant's fear, anxious, hyper arousal, and somatic symptoms pertaining to arousal. Items are normed to T-scores (mean = 50, standard deviation = 10), with higher T-scores indicating higher anxiety.
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 51 (10) | 52.9 (10.1)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 47.9 (10.2) | 53.7 (11)

21. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: Rate of a participant's pain experience, with items ranging from 0-4, and total scores ranging from 0-52, with higher scores indicating higher levels of pain catastrophizing
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline: number analyzed (Participants) | 9 | 10
  Baseline | 9.4 (6.8) | 11.6 (9.4)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 7.1 (5.6) | 11 (7.1)

22. Secondary Outcome: UCLA Loneliness Scale
Description: Rate of a participant's feelings of loneliness and social isolation and items range from 0-3, with a higher score reflecting greater feelings of loneliness, with total scores ranging from 0-24
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 12.9 (3.3) | 13.4 (4.4)
  Post-Test: number analyzed (Participants) | 8 | 9
  Post-Test | 12.6 (5.2) | 13.3 (3.6)

23. Secondary Outcome: Pain Self Efficacy Questionnaire (PSEQ)
Description: Rate of a participant's confidence to do various activities despite their pain, with items ranging from 0-6, and a higher score showing greater levels of confidence with pain self-efficacy, with total scores ranging from 0-60
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
score on a scale
  Baseline | 38 (14.2) | 35.5 (18.9)
  Post-Test: number analyzed (Participants) | 7 | 10
  Post-Test | 42.9 (14.5) | 38 (13.5)

24. Secondary Outcome: Tampa Kinesiophobia Scale
Description: Rate of a participant's fear of movement, with items ranging from 1-4, and a total scores ranging from 17-68, and higher scores indicating higher levels of fear of movement
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 8 | 9
score on a scale
  Baseline: number analyzed (Participants) | 8 | 8
  Baseline | 31.9 (6.2) | 37.6 (8.9)
  Post-Test: number analyzed (Participants) | 6 | 9
  Post-Test | 31.2 (13.5) | 35.8 (7.4)

25. Secondary Outcome: Chronic Pain Acceptance Questionnaire
Description: Rate of a participant's acceptance of chronic pain, with scores ranging from 0-6, with the total score ranging from 0-48, and higher scores indicating higher levels of acceptance of chronic pain
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 8 | 11
score on a scale
  Baseline | 30.1 (8.7) | 24.3 (10.7)
  Post-Test: number analyzed (Participants) | 7 | 11
  Post-Test | 31 (8.2) | 27.1 (3.7)

26. Secondary Outcome: Self-Compassion Scale (SCS)
Description: Rate of a participant's amount of self-compassion, with items ranging from 1-5, and total scores ranging from 12-60 and higher scores indicating higher levels of self-compassion
Time Frame: 0 Weeks, 8 Weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 8 | 11
score on a scale
  Baseline | 45.6 (7.9) | 44.4 (8.5)
  Post-Test: number analyzed (Participants) | 8 | 10
  Post-Test | 43.2 (7.4) | 43.6 (6.9)

27. Secondary Outcome: ActiGraph Average Steps
Description: Participants wore a ActiGraph accelerometer around their waist for 8 days to measure their daily average step count.
Time Frame: 0 weeks, 8 weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 10
steps per day
  Baseline: number analyzed (Participants) | 9 | 9
  Baseline | 3643.1 (1679.9) | 3195.3 (1975.7)
  Post-Test: number analyzed (Participants) | 8 | 10
  Post-Test | 4283.8 (1905.7) | 2604.4 (1912.8)

28. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: The Six-Minute Walk Test (6MWT) measures the distances participants can walk at an accelerated pace in meters over a 6-minute span.
Time Frame: 0 weeks, 8 weeks
Population: Participant dropout as cited in consort.
Measure: Mean (Standard Deviation); unit: meters per 6 minutes
Arm/Group | Active Brains | Active Brains 2
Number analyzed (Participants) | 9 | 11
meters per 6 minutes
  Baseline: number analyzed (Participants) | 9 | 10
  Baseline | 407.6 (110.2) | 415.6 (123.1)
  Post-Test: number analyzed (Participants) | 8 | 11
  Post-Test | 426.6 (147.6) | 435.2 (101.6)

ADVERSE EVENTS:
Time Frame: No adverse events required assessment at any point during the study period (1 year, 9 months).
Description: Because this is a behavioral intervention trial not requiring medication, there were no forseeable risks from participating in this research study. Thus, the number of participants at risk for Serious Adverse Events and All Cause Mortality was zero.
  We defined "Other" risks as feeling uncomfortable while completing various psychological questionnaires and possible discomfort with the topics of discussion in group sessions.
Arm/Group | Active Brains | Active Brains 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT04044183/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04044183/SAP_001.pdf